CLINICAL TRIAL: NCT07017075
Title: 3D Visulization The Area Of Maximal Compression And Quantitative Assessment Stroke Volume And Ejection Fraction After Adjusting CPR Location
Brief Title: Adjusting CPR Location With TEE Guidance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202410013RINB
Record Dates: First submitted 2025-05-06; First posted 2025-06-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest (CA)
Keywords: OHCA; TEE
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPR location without adjustment (Other): If the AMC was located at the LV identified by TEE, the CPR compression site was not altered.
  Interventions: Behavioral: adjustment of CPR location
- CPR location with adjustment (Other): If the AMC was not located at the LV, the CPR compression site was altered.
  Interventions: Behavioral: adjustment of CPR location

INTERVENTIONS:
Behavioral: adjustment of CPR location — Transesophageal ultrasound with built-in ultrasound software (Philips QLAB 3D quantification advance, Philips Healthcare, USA, speckle tracking echocardiography (STE,Speckle tracking echocardiography) to evaluate stroke volume and cardiac output in traditional CPR location and the better position

SUMMARY:
Use Transesophageal ultrasound in OHCA patients to identify the proper compression location

DETAILED DESCRIPTION:
For patients with cardiac arrest, high-quality cardiopulmonary resuscitation is performed according to critical care management and Advanced Cardiac Life Support (ACLS). Rapid with powerful chest compression should be performed to maintain the heart's output and blood flow. An advanced airway should be established and adjust resuscitation based on collected clinical information. Transesophageal ultrasound examination is performed after the advanced airway is established without affecting the resuscitation. The investigators use the built-in ultrasound software (Philips QLAB 3D quantification advance, Philips Healthcare, USA, speckle tracking echocardiography (STE,Speckle tracking echocardiography)) to analyze stroke volume and cardiac output. The investigators collect the stroke volume and cardiac output at the chest compression position recommended by ACLS, as well as the stroke volume and cardiac output after adjusting the optimal chest compression position. The investigators expect it can increase the return of spontaneous circulation rate, survival rate, and neurological prognosis over time.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest patients

Exclusion Criteria:

* DNR was signed
* Age under 18
* Trauma patients
* Patients hard to establish an advanced airway
* Inavailability of ultrasound machine or operators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
stroke volume, ejection fraction, end-diastolic volume, and end-systolic volume | 2 mins
  built-in ultrasound software (Philips QLAB 3D quantification advance, Philips Healthcare, USA, speckle tracking echocardiography (STE,Speckle tracking echocardiography)

CONTACTS AND LOCATIONS:
Overall Officials: WANCHING LIEN, Study Director — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Chang Bing Show Chawan Memorial Hospital, Changhua
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication

REFERENCES:
- [Result] Chen CC, Huang CS, Yen HT, Lien WC. A visualization of ejection fraction change after adjusting the area of maximal compression. Resuscitation. 2024 Jan;194:110097. doi: 10.1016/j.resuscitation.2023.110097. Epub 2023 Dec 20. No abstract available. PMID 38128870
- [Result] Teran F, Owyang CG, Martin-Flores M, Lao D, King A, Palasz J, Araos JD. Hemodynamic impact of chest compression location during cardiopulmonary resuscitation guided by transesophageal echocardiography. Crit Care. 2023 Aug 19;27(1):319. doi: 10.1186/s13054-023-04575-7. No abstract available. PMID 37598201
- [Result] Hwang SO, Zhao PG, Choi HJ, Park KH, Cha KC, Park SM, Kim SC, Kim H, Lee KH. Compression of the left ventricular outflow tract during cardiopulmonary resuscitation. Acad Emerg Med. 2009 Oct;16(10):928-33. doi: 10.1111/j.1553-2712.2009.00497.x. Epub 2009 Sep 3. PMID 19732038
- [Result] Olasveengen TM, Semeraro F, Ristagno G, Castren M, Handley A, Kuzovlev A, Monsieurs KG, Raffay V, Smyth M, Soar J, Svavarsdottir H, Perkins GD. European Resuscitation Council Guidelines 2021: Basic Life Support. Resuscitation. 2021 Apr;161:98-114. doi: 10.1016/j.resuscitation.2021.02.009. Epub 2021 Mar 24. PMID 33773835